CLINICAL TRIAL: NCT00420641
Title: A Ten-week, Multicenter, Randomized, Double-Blind, Placebo-and Active-Controlled, Paralleled-Group, Flexible-Dose Study Evaluating the Efficacy, Safety and Tolerability of GSK372475 or Paroxetine Compared to Placebo in Adult Subjects Diagnosed With Major Depressive Disorder
Brief Title: MDD POC Study GSK372475 Subjects Depressive Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SND 103288
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2014-10

CONDITIONS: Depressive Disorder
Keywords: MDD; flexible-dose; Major Depressive Disorder; paroxetine; GSK372475
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major | interventions — GSK372475; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK372475 Arm (Experimental): GSK372475 1.0- 1.5 mg/day
  Interventions: Drug: GSK372475
- Paroxetine Arm (Experimental): Paroxetine 20-30 mg/day
  Interventions: Drug: Paroxetine
- Placebo (Other): Placebo to Match
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSK372475 — GSK372475 1.0-1.5 mg/day
  Arms: GSK372475 Arm
Drug: Paroxetine — Paroxetine 20-30 mg/day
  Arms: Paroxetine Arm
Other: Placebo — Placebo to Match
  Arms: Placebo

SUMMARY:
To evaluate the efficacy, safety and tolerability of GSK372475 compared with placebo in the treatment of outpatients subjects with major depressive disorder to exhibit decreased pleasure, interest and energy.

ELIGIBILITY:
Inclusion criteria:

* Major depressive episode (MDE) associated with Major Depressive Disorder (DSM-IV-TR criteria)
* Duration of current episode is at least 12 weeks duration and less than 2 years
* Symptoms of decreased energy, pleasure, and interest
* Female subjects who agree to use acceptable methods of birth control throughout the study

Exclusion criteria:

* Current diagnosis of Panic Disorder, or symptoms of generalized anxiety or panic attacks that could interfere with their ability to complete the trial
* Symptoms of MDE better accounted for by another diagnosis
* Diagnosis of panic disorder / attacks, generalised anxiety, borderline or antisocial personality disorder, dementia, anorexia nervosa / bulimia (within 6 months of screening), bipolar disorder, schizophrenia or any other psychotic disorder(s).
* Started psychotherapy within 3 months prior to the Screening
* Received electroconvulsive therapy or transcranial magnetic stimulation within 6 months prior to screening
* Received psychoactive drugs within 4 weeks of randomization
* Positive urine drug screen or positive blood alcohol
* Suicidal risk or has had any previous suicide attempt, a family history of suicide attempt
* Positive pregnancy test
* History of seizure disorder, myocardial infarction (< 1yr), or unstable medical condition
* Failed to respond to an adequate course of pharmacotherapy of at least 2 different antidepressants

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 492 (Actual)
Dates: Start 2006-12-19; Primary Completion 2008-06-01 (Actual); Study Completion 2008-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Canada (4):
  - GSK Investigational Site, Miramichi, New Brunswick
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Markham, Ontario
  - GSK Investigational Site, Mississauga, Ontario
- Chile (2):
  - GSK Investigational Site, Providencia / Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Costa Rica (2):
  - GSK Investigational Site, Los Yoses, San José, Provincia de San José
  - GSK Investigational Site, San José
- Croatia (2):
  - GSK Investigational Site, Split
  - GSK Investigational Site, Zagreb
- France (5):
  - GSK Investigational Site, Angoulême
  - GSK Investigational Site, Dole
  - GSK Investigational Site, Élancourt
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Germany (4):
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Hüttenberg, Hesse
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin
- India (4):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Mangalore
  - GSK Investigational Site, Manipal
- Italy (2):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pisa, Tuscany
- Poland (3):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Chełmno
  - GSK Investigational Site, Leszno

REFERENCES:
- [Background] Learned S, Graff O, Roychowdhury S, Moate R, Krishnan KR, Archer G, Modell J, Alexander R, Zamuner S, Lavergne A, Evoniuk G, Ratti E. Results of Two Double-Blind, Placebo- and Active-Controlled Studies of GSK372475, a Triple Monoamine Reuptake Inhibitor, in the Treatment of Major Depressive Disorder. [J Psychopharmacol EPublication ahead of print. DOI 10.1177/0269881111424931]. 2011;
- [Derived] Learned S, Graff O, Roychowdhury S, Moate R, Krishnan KR, Archer G, Modell JG, Alexander R, Zamuner S, Lavergne A, Evoniuk G, Ratti E. Efficacy, safety, and tolerability of a triple reuptake inhibitor GSK372475 in the treatment of patients with major depressive disorder: two randomized, placebo- and active-controlled clinical trials. J Psychopharmacol. 2012 May;26(5):653-62. doi: 10.1177/0269881111424931. Epub 2011 Nov 2. PMID 22048884

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted on male and female participants, aged 18 to 64, with major depressive episodes associated with major depressive disorder (MDD), from 19 December 2006 to 24 June 2008 at 35 centers in 10 countries of Canada (4), Bulgaria (2), Croatia (5), France (4), Germany (4), Italy (2), Poland (3), Chile (3), Costa Rica (3) and India (5).
Pre-assignment Details: A total of 504 participants were randomized in ratio of 1:1:1 to receive placebo or GSK372475 (1.0 milligram per day [mg/day] to 1.5 mg/day) or paroxetine (20 mg/day to 30 mg/day) for 10 week double blind treatment phase.
Groups:
- Placebo: Participants received oral dose of matching placebo to capsule GSK372475/paroxetine for dose level 1 (DL1) once daily in morning for 4 weeks of treatment period and DL2 once daily in morning for remaining 6 weeks. Dose escalation was based on investigator's judgement of participant not experiencing any troublesome adverse signs or symptoms and not meeting response criteria (>=50% reduction from randomization in Montgomery-Asberg Depression Rating Scale [MADRS] total score). Treatment Phase of study was followed by a one week Taper Phase where participants were dosed placebo capsules to maintain blind for Taper Phase of paroxetine, applicable for all participants who completed 10 week double-blind treatment phase on DL2 or who withdrew prematurely after having received at least 1 week of study medication on DL2. Lorazepam (or other specified comparable sedative) was permitted as a night-time sleep aid at the recommended dosage during first 2 weeks of study starting at randomization.
- GSK372475: Participants received oral dose of GSK372475 1.0 mg/day capsule at dose level 1 (DL1) once daily in morning for 4 weeks of treatment period and 1.5 mg/day capsule once daily in morning at DL2 for remaining 6 weeks. Dose escalation was based on investigator's judgement of participant not experiencing any troublesome adverse signs or symptoms and not meeting response criteria (>=50% reduction from randomization in MADRS total score). Treatment Phase of study was followed by a one week Taper Phase where participants were dosed placebo capsules to maintain blind for Taper Phase of paroxetine, applicable for all participants who completed 10 week double-blind treatment phase on DL2 or who withdrew prematurely after having received at least 1 week of study medication on DL2. Lorazepam (or other specified comparable sedative) was permitted as a night-time sleep aid at the recommended dosage during first 2 weeks of study starting at randomization.
- Paroxetine: Participants received oral dose of paroxetine 20 mg/day capsule at DL1 once daily in morning for 4 weeks of treatment period and 30 mg/day capsule once daily in morning at DL2 for remaining 6 weeks. Dose escalation was based on the investigator's judgement of participant not experiencing any troublesome adverse signs or symptoms and not meeting response criteria (>=50% reduction from randomization in MADRS total score). Treatment Phase of study was followed by a one week Taper Phase where participants were dosed at DL1, applicable for all participants who completed 10 week double-blind treatment phase on DL2 or who withdrew prematurely after having received at least 1 week of study medication on DL2. Lorazepam (or other specified comparable sedative) was permitted as a night-time sleep aid at the recommended dosage during first 2 weeks of study starting at randomization.
Period: Overall Study
Arm/Group | Placebo | GSK372475 | Paroxetine
Started | 160 | 172 | 172
Completed | 115 | 100 | 128
Not Completed | 45 | 72 | 44
Not completed — Adverse Event | 3 | 25 | 10
Not completed — Lost to Follow-up | 2 | 4 | 2
Not completed — Protocol Violation | 8 | 8 | 7
Not completed — Withdrawal by Subject | 15 | 21 | 14
Not completed — Lack of Efficacy | 6 | 5 | 4
Not completed — Non-compliance | 7 | 5 | 4
Not completed — Other | 4 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population was defined as consisting of all participants who gave informed consent, were randomized, received at least one dose of double blind medication and for whom at least one post-randomization assessment was available.
Groups:
- Placebo: Participants received oral dose of matching placebo to capsule GSK372475/paroxetine for DL1 once daily in morning for 4 weeks of treatment period and DL2 once daily in morning for remaining 6 weeks. Dose escalation was based on investigator's judgement of participant not experiencing any troublesome adverse signs or symptoms and not meeting response criteria (>=50% reduction from randomization in MADRS total score). Treatment Phase of study was followed by a one week Taper Phase where participants were dosed placebo capsules to maintain blind for Taper Phase of paroxetine, applicable for all participants who completed 10 week double-blind treatment phase on DL2 or who withdrew prematurely after having received at least 1 week of study medication on DL2. Lorazepam (or other specified comparable sedative) was permitted as a night-time sleep aid at the recommended dosage during first 2 weeks of study starting at randomization.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK372475 | Paroxetine | Total
Number analyzed (Participants) | 156 | 171 | 166 | 493
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (10.89) | 42.4 (11.64) | 44.4 (10.90) | 42.9 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 117 | 111 | 345
  Male | 39 | 54 | 55 | 148
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant in the placebo arm did not have any data recorded for geographic ancestry. However the investigator commented that the participant was 'West Indian'.
  Participants
    number analyzed (Participants) | 155 | 171 | 166 | 492
    American Indian or Alaska Native | 8 | 11 | 11 | 30
    Asian | 13 | 14 | 12 | 39
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
    Black or African American | 2 | 0 | 2 | 4
    White | 128 | 144 | 137 | 409
    More than one race | 3 | 2 | 4 | 9
    Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Randomization at the End of the Treatment Phase in the MADRS Total Score
Description: The MADRS scale measures the depression level of a participant. The total score was derived by adding the scores of the following 10 items: 1, apparent sadness; 2, reported sadness; 3, inner tension; 4, reduced sleep; 5, reduced appetite; 6, concentration difficulties; 7, lassitude; 8, inability to feel; 9, pessimistic thoughts; 10, suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). The maximum total score is 60; 0, no depression; 60, severely depressed. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between MADRS total score at the time point being analyzed (Week 10) to Randomization.
Time Frame: Week 0 (Randomization) and Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 117 | 100 | 130
Score on scale | -16.9 (9.97) | -19.0 (9.50) | -20.5 (8.65)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS total score at Week 10; Test type: Superiority or Other; p = 0.485, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = -0.78, 90% CI 2-sided [-2.60 to 1.05] — The point estimate was calculated as least square (LS) mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS total score at Week 10; Test type: Superiority or Other; p = 0.000, MMRM; Mean Difference (Final Values) = -3.99, 90% CI 2-sided [-5.75 to -2.22] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

2. Primary Outcome: Change From Randomization at the End of the Treatment Phase (Week 10) in Bech Scale (6-item of 17-item Hamilton Depression Rating [HAMD-17] Scale) Score
Description: The HAMD is a rating instrument for evaluating severity of symptoms of depression, was completed by the participant. The rating instrument used in this study was the 17-item version (HAM-D17). The Bech scale of the HAMD-17 is composed of 6 identified items out of the 17 items rated in HAMD-17 scale. Each item is rated on either a 3-point scale (0 to 2) or a 5-point scale (0 to 4). The following symptoms were rated on a 5-point scale (0-4): depressed mood, feeling of guilt, work and interests, psychomotor retardation, and anxiety (psychic). The following symptom was rated on a 3-point scale (0-2): somatic symptoms (general). Total score ranged from 0 to 22, with 0 indicating absence of symptoms and a higher score indicating greater severity of symptoms. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between Bech total score at the time point being analyzed (Week 10) to Randomization.
Time Frame: Week 0 (Randomization) and Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 117 | 100 | 130
Score on scale | -6.2 (4.32) | -7.2 (3.98) | -7.9 (3.82)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in Bech score at Week 10; Test type: Superiority or Other; p = 0.252, MMRM; Mean Difference (Final Values) = -0.53, 90% CI 2-sided [-1.28 to 0.23] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS total score at Week 10; Test type: Superiority or Other; p = 0.000, MMRM; Mean Difference (Final Values) = -1.77, 90% CI 2-sided [-2.49 to -1.05] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

3. Primary Outcome: Mean Change From Randomization at the End of the Treatment Phase (Week 10) in Inventory of Depressive Symptomatology-Clinician Rated (IDS-CR) Total Score
Description: The IDS-CR is a standardized 30-item, clinician rated scale to assess the severity of a participant's depressive symptoms. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. In order to calculate the total score of IDS-CR, the following procedures were used: either item 11 or 12 were scored; either item 13 or 14 were scored; if both items 11 and 12 (or 13 and 14) were scored, the highest of the items was scored. The total score was obtained by adding the scores of 28 items of the 30 items. Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between IDS-CR total score at the time point being analyzed (Week 10) to Randomization.
Time Frame: Week 0 (Randomization) and Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 117 | 100 | 130
Score on scale | -22.3 (14.21) | -25.1 (13.30) | -26.8 (12.10)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR total score at Week 10; Test type: Superiority or Other; p = 0.279, MMRM; Mean Difference (Final Values) = -1.66, 90% CI 2-sided [-4.19 to 0.87] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR total score at Week 10; Test type: Superiority or Other; p = 0.001, MMRM; Mean Difference (Final Values) = -5.12, 90% CI 2-sided [-7.55 to -2.68] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

4. Secondary Outcome: Mean Change From Randomization in IDS- Self-Rated Version (SR) Total Score Over Week 10
Description: The IDS-SR is a standardized 30-item, participant rated scale to assess the severity of a participant's depressive symptoms. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. In order to calculate the total score of IDS-SR, the following procedures were used: either item 11 or 12 were scored; either item 13 or 14 were scored; if both items 11 and 12 (or 13 and 14) were scored, the highest of the items was scored. The total score was obtained by adding the scores of 28 items of the 30 items. Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between IDS-SR total score at the individual time points being analyzed (Week, 1, 4 and 10) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 132 | 144 | 151
  Week 1 | -7.6 (9.05) | -7.6 (9.15) | -8.6 (9.96)
  Week 4: number analyzed (Participants) | 119 | 119 | 122
  Week 4 | -16.8 (12.12) | -15.5 (13.00) | -19.1 (12.55)
  Week 10: number analyzed (Participants) | 103 | 89 | 117
  Week 10 | -25.6 (16.27) | -26.9 (14.73) | -30.5 (13.66)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-SR total score at Week 10; Test type: Superiority or Other; p = 0.287, MMRM; Mean Difference (Final Values) = -2.05, 90% CI 2-sided [-5.23 to 1.12] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-SR total score at Week 10; Test type: Superiority or Other; p = 0.001, MMRM; Mean Difference (Final Values) = -6.23, 90% CI 2-sided [-9.21 to -3.25] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

5. Secondary Outcome: Mean Change From Randomization in the 16-item Quick Inventory of Depressive Symptomatology-Clinician-rated Version (QIDS-CR16) Total Score Over Week 10
Description: QIDS-CR16 is a 16-item rating scale of depressive symptoms rated by the clinician. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Total score was obtained by adding scores of items of sad mood, interest, energy/fatigue, sleep disturbance, decrease/increase in appetite or weight, concentration/decision making, suicidal ideation and psychomotor agitation/retardation, the highest score on any 1 of the 4 sleep items, highest score on any 1 appetite/weight item and highest score on either of the 2 psychomotor items. Total scores range from 0-27, with a score of 0 indicating no depression and a score of 27 indicating most severe depression. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between QIDS-CR16 total score at the individual time points being analyzed (Week 1, 2, 3, 4, 5, 6, 8 and 10) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 150 | 167 | 164
  Week 1 | -1.5 (2.78) | -1.8 (2.76) | -1.8 (3.65)
  Week 2: number analyzed (Participants) | 145 | 151 | 152
  Week 2 | -3.3 (3.67) | -3.6 (4.01) | -3.4 (4.70)
  Week 3: number analyzed (Participants) | 137 | 144 | 151
  Week 3 | -5.0 (4.27) | -4.3 (4.24) | -5.3 (4.64)
  Week 4: number analyzed (Participants) | 138 | 138 | 147
  Week 4 | -5.9 (4.75) | -5.0 (4.20) | -5.9 (4.61)
  Week 5: number analyzed (Participants) | 128 | 123 | 140
  Week 5 | -6.5 (4.64) | -6.6 (5.09) | -7.4 (4.82)
  Week 6: number analyzed (Participants) | 129 | 116 | 136
  Week 6 | -7.3 (4.88) | -7.3 (5.55) | -8.6 (4.92)
  Week 8: number analyzed (Participants) | 116 | 103 | 133
  Week 8 | -7.8 (5.58) | -8.8 (5.07) | -9.4 (5.03)
  Week 10: number analyzed (Participants) | 117 | 100 | 130
  Week 10 | -8.5 (5.31) | -9.6 (4.95) | -10.0 (4.85)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in QIDS-CR16 total score at Week 10; Test type: Superiority or Other; p = 0.352, MMRM; Mean Difference (Final Values) = -0.53, 90% CI 2-sided [-1.47 to 0.41] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in QIDS-CR16 total score at Week 10; Test type: Superiority or Other; p = 0.002, MMRM; Mean Difference (Final Values) = -1.71, 90% CI 2-sided [-2.62 to -0.81] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

6. Secondary Outcome: Mean Change From Randomization in the 16-item Quick Inventory of Depressive Symptomatology-Self-rated Version (QIDS-SR16) Total Score Over Week 10
Description: QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by participant. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Total score was obtained by adding scores of the items of sad mood, interest, energy/fatigue, sleep disturbance, decrease/increase in appetite or weight, concentration/decision making, suicidal ideation and psychomotor agitation/retardation, the highest score on any 1 of the 4 sleep items, highest score on any 1 appetite/weight item and highest score on either of the 2 psychomotor items. Total scores range from 0-27, with a score of 0 indicating no depression and a score of 27 indicating most severe depression. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between QIDS-SR16 total score at the individual time points being analyzed (Week 1, 4 and 10) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 130 | 141 | 151
  Week 1 | -2.7 (3.82) | -3.1 (4.00) | -2.9 (4.16)
  Week 4: number analyzed (Participants) | 118 | 119 | 122
  Week 4 | -6.4 (5.23) | -5.7 (5.31) | -6.9 (5.10)
  Week 10: number analyzed (Participants) | 102 | 89 | 117
  Week 10 | -10.0 (6.73) | -10.6 (5.64) | -11.6 (5.39)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in QIDS-SR16 total score at Week 10; Test type: Superiority or Other; p = 0.168, MMRM; Mean Difference (Final Values) = -1.03, 90% CI 2-sided [-2.27 to 0.20] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in QIDS-SR16 total score at Week 10; Test type: Superiority or Other; p = 0.002, MMRM; Mean Difference (Final Values) = -2.12, 90% CI 2-sided [-3.27 to -0.97] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

7. Secondary Outcome: Mean Change From Randomization in the MADRS Item 2 Score (Reported Sadness) Over Week 10
Description: The MADRS scale measures the depression level of a participant. The items of the scale include: 1, apparent sadness; 2, reported sadness; 3, inner tension; 4, reduced sleep; 5, reduced appetite; 6, concentration difficulties; 7, lassitude; 8, inability to feel; 9, pessimistic thoughts; 10, suicidal thoughts. The item 2 (Reported Sadness) of MADRS was scored using a scale 7-point scale of 0-6, where 0 indicates absence of symptom and higher score indicates increased severity of symptom. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between MADRS Item 2 score at the time points being analyzed (Week 1, 2, 3, 4, 5, 6, 8 and 10) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 150 | 167 | 164
  Week 1 | -0.4 (0.84) | -0.5 (0.95) | -0.4 (0.97)
  Week 2: number analyzed (Participants) | 145 | 151 | 152
  Week 2 | -0.8 (1.00) | -0.9 (1.15) | -0.9 (1.27)
  Week 3: number analyzed (Participants) | 137 | 144 | 151
  Week 3 | -1.3 (1.26) | -1.2 (1.28) | -1.5 (1.28)
  Week 4: number analyzed (Participants) | 138 | 138 | 147
  Week 4 | -1.5 (1.42) | -1.4 (1.23) | -1.6 (1.34)
  Week 5: number analyzed (Participants) | 128 | 123 | 140
  Week 5 | -1.6 (1.43) | -1.7 (1.42) | -2.1 (1.28)
  Week 6: number analyzed (Participants) | 129 | 116 | 136
  Week 6 | -1.9 (1.56) | -2.0 (1.53) | -2.4 (1.29)
  Week 8: number analyzed (Participants) | 116 | 103 | 133
  Week 8 | -2.0 (1.43) | -2.4 (1.33) | -2.6 (1.34)
  Week 10: number analyzed (Participants) | 117 | 100 | 130
  Week 10 | -2.4 (1.52) | -2.7 (1.36) | -2.9 (1.28)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS Item 2 score at Week 10; Test type: Superiority or Other; p = 0.257, MMRM; Mean Difference (Final Values) = -0.19, 90% CI 2-sided [-0.46 to 0.09] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS Item 2 score at Week 10; Test type: Superiority or Other; p = 0.001, MMRM; Mean Difference (Final Values) = -0.51, 90% CI 2-sided [-0.77 to -0.25] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

8. Secondary Outcome: Mean Change From Randomization in the IDS-CR Scale Item 5 (Feeling Sad) Over Week 10
Description: The IDS-CR is a standardized 30-item, clinician rated scale to assess the severity of a participant's depressive symptoms. The item 5 (Feeling Sad) of IDS-CR was rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in score was the difference between IDS-CR Item 5 score at the time points being analyzed (Week 1, 2, 3, 4, 5, 6, 8 and 10) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 150 | 167 | 164
  Week 1 | -0.2 (0.61) | -0.3 (0.70) | -0.3 (0.75)
  Week 2: number analyzed (Participants) | 145 | 151 | 152
  Week 2 | -0.5 (0.72) | -0.5 (0.85) | -0.6 (0.87)
  Week 3: number analyzed (Participants) | 137 | 144 | 151
  Week 3 | -0.8 (0.74) | -0.8 (0.91) | -0.9 (0.82)
  Week 4: number analyzed (Participants) | 138 | 138 | 147
  Week 4 | -0.9 (0.84) | -0.8 (0.93) | -1.0 (0.83)
  Week 5: number analyzed (Participants) | 128 | 123 | 140
  Week 5 | -1.0 (0.84) | -1.0 (1.06) | -1.3 (0.86)
  Week 6: number analyzed (Participants) | 129 | 116 | 136
  Week 6 | -1.1 (0.90) | -1.2 (1.12) | -1.5 (0.87)
  Week 8: number analyzed (Participants) | 116 | 103 | 133
  Week 8 | -1.2 (0.92) | -1.4 (0.98) | -1.6 (0.90)
  Week 10: number analyzed (Participants) | 117 | 100 | 130
  Week 10 | -1.3 (0.95) | -1.5 (0.99) | -1.7 (0.88)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR Item 5 score at Week 10; Test type: Superiority or Other; p = 0.096, MMRM; Mean Difference (Final Values) = -0.17, 90% CI 2-sided [-0.33 to -0.00] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR Item 5 at Week 10; Test type: Superiority or Other; p = 0.000, MMRM; Mean Difference (Final Values) = -0.37, 90% CI 2-sided [-0.53 to -0.22] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

9. Secondary Outcome: Mean Change From Randomization at the End of the Treatment Phase (Week 10) in the HAMD-17 Total Score
Description: HAMD-17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items of HAMD-17 are rated on a scale 3-point scale of 0-2 or a 5-point scale of 0-4 where 0 is absence of symptom and higher score indicate more severe symptom. Items rated on the 3-point scale include: insomnia early, middle, late; somatic symptoms gastrointestinal and general; genital symptoms; loss of weight; insight. Items rated on 5-point scale include: depressed mood; feelings of guilt; suicide; work and activities; retardation; agitation; anxiety psychic and somatic; hypochondriasis. Total score ranges from 0 to 52, where 0 indicates absence of symptom and higher scores indicates more severe symptoms. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between HAMD-17 total score at the time point being analyzed (Week 10) to Randomization.
Time Frame: Week 0 (Randomization) and Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 150 | 167 | 164
  Week 1 | -1.9 (4.11) | -1.9 (4.16) | -2.3 (4.36)
  Week 2: number analyzed (Participants) | 145 | 151 | 152
  Week 2 | -4.3 (4.87) | -4.2 (5.82) | -4.8 (5.99)
  Week 3: number analyzed (Participants) | 137 | 144 | 151
  Week 3 | -6.6 (5.66) | -4.9 (6.73) | -6.9 (6.39)
  Week 4: number analyzed (Participants) | 138 | 138 | 147
  Week 4 | -7.7 (6.51) | -6.3 (6.30) | -7.9 (6.43)
  Week 5: number analyzed (Participants) | 128 | 123 | 140
  Week 5 | -8.5 (6.36) | -7.8 (7.68) | -9.9 (6.34)
  Week 6: number analyzed (Participants) | 129 | 116 | 136
  Week 6 | -9.9 (7.08) | -9.5 (8.38) | -11.6 (6.62)
  Week 8: number analyzed (Participants) | 116 | 103 | 133
  Week 8 | -10.4 (7.88) | -11.5 (7.78) | -12.7 (7.02)
  Week 10: number analyzed (Participants) | 117 | 100 | 130
  Week 10 | -11.5 (7.73) | -12.9 (7.46) | -13.9 (6.89)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 total score at Week 10; Test type: Superiority or Other; p = 0.576, MMRM; Mean Difference (Final Values) = -0.47, 90% CI 2-sided [-1.84 to 0.91] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 total score at Week 10; Test type: Superiority or Other; p = 0.000, MMRM; Mean Difference (Final Values) = -2.96, 90% CI 2-sided [-4.28 to -1.64] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

10. Secondary Outcome: Mean Change From Randomization in the HAMD-17 Scale Item 1 (Depressed Mood) Over Week 10
Description: HAMD-17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, work and activities, sleep, suicide, psychomotor agitation/retardation, appetite, sexual interest, anxiety, and somatic symptoms). The items of the HAMD-17 are rated on a 3-point scale of 0-2 or a 5-point scale of 0-4. The item 1 (Depressed Mood) of HAMD-17 was rated the 5-point scale of 0-4, where 0 indicates absence of symptom and higher score indicates more severe symptom. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in the score was the difference between HAMD-17 Item 1 score at the individual time points being analyzed (Week 1, 2, 3, 4, 5, 6, 8 and 10) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 10
Population: ITT Population with OC analysis. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 150 | 167 | 164
  Week 1 | -0.3 (0.69) | -0.4 (0.83) | -0.3 (0.79)
  Week 2: number analyzed (Participants) | 145 | 151 | 152
  Week 2 | -0.6 (0.84) | -0.7 (1.03) | -0.7 (0.97)
  Week 3: number analyzed (Participants) | 137 | 144 | 151
  Week 3 | -1.0 (1.06) | -0.9 (1.12) | -1.0 (1.01)
  Week 4: number analyzed (Participants) | 138 | 138 | 147
  Week 4 | -1.0 (1.10) | -1.0 (1.10) | -1.2 (1.04)
  Week 5: number analyzed (Participants) | 128 | 123 | 140
  Week 5 | -1.2 (1.11) | -1.2 (1.21) | -1.5 (1.06)
  Week 6: number analyzed (Participants) | 129 | 116 | 136
  Week 6 | -1.3 (1.16) | -1.5 (1.31) | -1.7 (1.03)
  Week 8: number analyzed (Participants) | 116 | 103 | 133
  Week 8 | -1.4 (1.18) | -1.8 (1.13) | -1.8 (1.06)
  Week 10: number analyzed (Participants) | 117 | 100 | 130
  Week 10 | -1.7 (1.24) | -2.0 (1.18) | -2.0 (1.06)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 Item 1 score at Week 10; Test type: Superiority or Other; p = 0.209, MMRM; Mean Difference (Final Values) = -0.16, 90% CI 2-sided [-0.38 to 0.05] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 Item 1 score at Week 10; Test type: Superiority or Other; p = 0.002, MMRM; Mean Difference (Final Values) = -0.39, 90% CI 2-sided [-0.60 to -0.19] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

11. Secondary Outcome: Mean Change From Randomization in IDS-CR and IDS-SR 5 Item Subscale Over Week 10
Description: The IDS-CR and IDS-SR is a standardized 30-item scale rated by the clinician and the participant respectively to assess the severity of a participant's depressive symptoms. The 5 items of the IDS subscale include: item 19 (general interest/involvement), item 20 (energy/fatigability), item 21 (pleasure/enjoyment), item 22 (sexual interest), item 30 (Leaden paralysis/physical energy) which assessed participant's pleasure, interest and energy. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Total score ranges from 0 to 15, where 0 indicates absence of symptom and higher scores indicates more severe symptoms. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between IDS 5 Item subscale total score at the individual time points being analyzed (Week 1, 2, 3, 4, 5, 6, 8 and 10) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  IDS-CR 5 Item subscale, Week 1: number analyzed (Participants) | 150 | 167 | 164
  IDS-CR 5 Item subscale, Week 1 | -0.8 (2.08) | -1.2 (2.32) | -0.8 (2.21)
  IDS-CR 5 Item subscale, Week 2: number analyzed (Participants) | 145 | 151 | 152
  IDS-CR 5 Item subscale, Week 2 | -1.6 (2.49) | -2.5 (2.85) | -2.0 (2.85)
  IDS-CR 5 Item subscale, Week 3: number analyzed (Participants) | 137 | 144 | 151
  IDS-CR 5 Item subscale, Week 3 | -2.6 (3.05) | -2.9 (3.13) | -2.9 (3.12)
  IDS-CR 5 Item subscale, Week 4: number analyzed (Participants) | 138 | 138 | 147
  IDS-CR 5 Item subscale, Week 4 | -3.1 (3.41) | -3.5 (3.13) | -3.4 (3.06)
  IDS-CR 5 Item subscale, Week 5: number analyzed (Participants) | 128 | 123 | 140
  IDS-CR 5 Item subscale, Week 5 | -3.8 (3.24) | -4.3 (3.60) | -4.4 (3.41)
  IDS-CR 5 Item subscale, Week 6: number analyzed (Participants) | 129 | 116 | 136
  IDS-CR 5 Item subscale, Week 6 | -4.4 (3.76) | -4.8 (3.81) | -5.2 (3.59)
  IDS-CR 5 Item subscale, Week 8: number analyzed (Participants) | 116 | 103 | 133
  IDS-CR 5 Item subscale, Week 8 | -4.8 (3.85) | -5.6 (3.56) | -5.9 (3.41)
  IDS-CR 5 Item subscale, Week 10: number analyzed (Participants) | 117 | 100 | 130
  IDS-CR 5 Item subscale, Week 10 | -5.3 (3.73) | -6.2 (3.42) | -6.3 (3.21)
  IDS-SR 5 Item subscale, Week 1: number analyzed (Participants) | 130 | 141 | 151
  IDS-SR 5 Item subscale, Week 1 | -1.3 (2.48) | -2.5 (3.10) | -2.2 (3.09)
  IDS-SR 5 Item subscale, Week 2: number analyzed (Participants) | 4 | 7 | 3
  IDS-SR 5 Item subscale, Week 2 | -3.0 (4.55) | -2.1 (2.97) | -3.3 (4.16)
  IDS-SR 5 Item subscale, Week 3: number analyzed (Participants) | 2 | 7 | 7
  IDS-SR 5 Item subscale, Week 3 | 0.0 (0.00) | -3.4 (5.91) | -3.7 (5.99)
  IDS-SR 5 Item subscale, Week 4: number analyzed (Participants) | 118 | 119 | 122
  IDS-SR 5 Item subscale, Week 4 | -3.5 (3.96) | -4.7 (4.12) | -4.9 (3.85)
  IDS-SR 5 Item subscale, Week 5: number analyzed (Participants) | 7 | 11 | 5
  IDS-SR 5 Item subscale, Week 5 | -0.7 (1.50) | -5.9 (3.81) | -5.0 (6.52)
  IDS-SR 5 Item subscale, Week 6: number analyzed (Participants) | 6 | 6 | 3
  IDS-SR 5 Item subscale, Week 6 | -2.8 (3.76) | -1.0 (5.37) | -3.3 (2.52)
  IDS-SR 5 Item subscale, Week 8: number analyzed (Participants) | 2 | 3 | 3
  IDS-SR 5 Item subscale, Week 8 | -2.5 (2.12) | -7.0 (3.61) | -6.3 (4.04)
  IDS-SR 5 Item subscale, Week 10: number analyzed (Participants) | 102 | 89 | 117
  IDS-SR 5 Item subscale, Week 10 | -6.2 (4.53) | -7.6 (4.21) | -7.9 (4.26)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR 5 Item subscale total score at Week 10; Test type: Superiority or Other; p = 0.175, MMRM; Mean Difference (Final Values) = -0.55, 90% CI 2-sided [-1.23 to 0.12] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR 5 Item subscale total score at Week 10; Test type: Superiority or Other; p = 0.003, MMRM; Mean Difference (Final Values) = -1.15, 90% CI 2-sided [-1.79 to -0.50] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine
Statistical Analysis 3: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-SR 5 Item subscale total score at Week 10; Test type: Superiority or Other; p = 0.082, MMRM; Mean Difference (Final Values) = -0.99, 90% CI 2-sided [-1.92 to -0.05] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 4: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-SR 5 Item subscale total score at Week 10; Test type: Superiority or Other; p = 0.001, MMRM; Mean Difference (Final Values) = -1.77, 90% CI 2-sided [-2.64 to -0.90] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

12. Secondary Outcome: Mean Change From Randomization in the Clinical Global Impression-Severity of Illness (CGI-S) Scale Over Week 10
Description: The CGI-S scale measures the severity of psychiatric symptoms on a 7-point scale from 1-7. The scores indicated the following: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants. The score ranged from 1-7, where 1 indicated absence of symptoms and higher score indicated greater severity of symptoms. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in the score was the difference between CGI-S score at the individual time points being analyzed (Week 1, 2, 3, 4, 5, 6, 8 and 10) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 10
Population: ITT Population with OC analysis. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 150 | 169 | 166
  Week 1 | -0.2 (0.54) | -0.3 (0.55) | -0.2 (0.56)
  Week 2: number analyzed (Participants) | 146 | 154 | 155
  Week 2 | -0.5 (0.70) | -0.5 (0.93) | -0.6 (0.88)
  Week 3: number analyzed (Participants) | 138 | 146 | 154
  Week 3 | -0.8 (0.91) | -0.7 (1.09) | -1.1 (1.19)
  Week 4: number analyzed (Participants) | 144 | 138 | 149
  Week 4 | -1.1 (1.11) | -1.0 (1.20) | -1.3 (1.28)
  Week 5: number analyzed (Participants) | 129 | 123 | 142
  Week 5 | -1.2 (1.23) | -1.4 (1.41) | -1.6 (1.28)
  Week 6: number analyzed (Participants) | 132 | 124 | 137
  Week 6 | -1.5 (1.30) | -1.6 (1.54) | -2.0 (1.36)
  Week 8: number analyzed (Participants) | 117 | 107 | 132
  Week 8 | -1.7 (1.40) | -1.9 (1.51) | -2.2 (1.31)
  Week 10: number analyzed (Participants) | 120 | 102 | 132
  Week 10 | -1.9 (1.41) | -2.2 (1.54) | -2.5 (1.27)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in CGI-S score at Week 10; Test type: Superiority or Other; p = 0.208, MMRM; Mean Difference (Final Values) = -0.19, 90% CI 2-sided [-0.45 to 0.06] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in CGI-S score at Week 10; Test type: Superiority or Other; p = 0.000, MMRM; Mean Difference (Final Values) = -0.52, 90% CI 2-sided [-0.76 to -0.28] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

13. Secondary Outcome: Mean Change From Randomization in the Motivation and Energy Inventory (MEI) 18-Item Short Form (SF) Total Score Over Week 10
Description: MEI 18 item-SF questionnaire was used to measure reductions in mental energy, physical energy, and social motivation. All items use either a 7-level (0-6) or 5-level (0-4) response scale; for questions 1, 2, and 13-18, response '0' indicates lower motivation, energy and interest and responses with higher scores indicate increased motivation, energy and interest. For questions 3-12, response '0' indicates higher motivation, energy and interest and responses with higher scores indicate lower motivation, energy and interest. Items with a 5-level response scale were rescaled to 7-levels, and items were reverse-scored. Total score ranges from 0-108, where 0 indicates lower motivation, energy and interest and higher score indicates higher motivation, energy and interest. Randomization value was defined as assessment value done on Week 0. Change from Randomization in total score was difference between MEI score at individual time points being analyzed (Week 1, 4 and 10) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 150 | 166 | 164
  Week 1 | 3.8 (10.18) | 5.7 (12.23) | 4.9 (12.02)
  Week 4: number analyzed (Participants) | 137 | 134 | 143
  Week 4 | 16.1 (16.18) | 15.4 (17.68) | 18.4 (18.14)
  Week 10: number analyzed (Participants) | 117 | 98 | 130
  Week 10 | 29.8 (23.46) | 31.8 (23.25) | 34.3 (21.07)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MEI total score at Week 10; Test type: Superiority or Other; p = 0.516, MMRM; Mean Difference (Final Values) = 1.76, 90% CI 2-sided [-2.71 to 6.24] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MEI total score at Week 10; Test type: Superiority or Other; p = 0.016, MMRM; Mean Difference (Final Values) = 6.22, 90% CI 2-sided [1.97 to 10.48] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

14. Secondary Outcome: Mean Change From Randomization in the Changes in Sexual Functioning Questionnaire 14-item Short Form (CSFQ-14SF) Over Week 10
Description: The CSFQ-14SF is a structured self reported questionnaire designed to measure illness- and medication-related changes in sexual functioning. It is consisting of 14 items that measure sexual activity and sexual functioning. It measures five dimensions of sexual behavior: pleasure (1 item); desire/frequency (items 2 and 3); desire/interest (items 4, 5 and 6); arousal (items 7, 8 and 9); and orgasm (items 11, 12 and 13). Items 10 and 14 are included in the total score but not in any dimension score. Items were rated on an 5 point scale from 1 to 5. Total score ranged from 14 to 70, where higher scores indicate higher sexual functioning and lower score indicate lower sexual functioning. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in the total score was the difference between CSFQ-14SF score at the individual time points being analyzed (Week 4 and 10) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 4: number analyzed (Participants) | 134 | 133 | 141
  Week 4 | 2.4 (5.44) | 3.1 (7.63) | 1.3 (8.08)
  Week 10: number analyzed (Participants) | 114 | 99 | 125
  Week 10 | 4.6 (8.17) | 6.1 (8.95) | 4.4 (9.30)
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in CSFQ-14SF total score at Week 10; Test type: Superiority or Other; p = 0.126, MMRM; Mean Difference (Final Values) = 1.72, 90% CI 2-sided [-0.13 to 3.57] — The point estimate was calculated as LS mean difference (final value) of placebo and GSK372475
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in CSFQ-14SF total score at Week 10; Test type: Superiority or Other; p = 0.957, MMRM; Mean Difference (Final Values) = 0.06, 90% CI 2-sided [-1.69 to 1.81] — The point estimate was calculated as LS mean difference (final value) of placebo and Paroxetine

15. Secondary Outcome: Mean Change From Randomization in the MADRS Total Score Over Week 8
Description: The MADRS scale measures the depression level of a participant. The total score was derived by adding the scores of the following 10 items: 1, apparent sadness; 2, reported sadness; 3, inner tension; 4, reduced sleep; 5, reduced appetite; 6, concentration difficulties; 7, lassitude; 8, inability to feel; 9, pessimistic thoughts; 10, suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). The total score ranged from 0-60, where 0 indicated no depression and 60 indicated severely depressed. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between MADRS total score at the time points being analyzed (Week 1, 2, 3, 4, 5, 6 and 8) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 150 | 167 | 164
  Week 1 | -2.9 (5.40) | -2.8 (5.61) | -2.8 (5.98)
  Week 2: number analyzed (Participants) | 145 | 151 | 152
  Week 2 | -6.3 (6.78) | -5.7 (7.62) | -6.6 (8.50)
  Week 3: number analyzed (Participants) | 137 | 144 | 151
  Week 3 | -9.7 (8.45) | -7.3 (8.56) | -10.1 (8.59)
  Week 4: number analyzed (Participants) | 138 | 138 | 147
  Week 4 | -11.0 (9.23) | -9.5 (8.08) | -11.4 (8.67)
  Week 5: number analyzed (Participants) | 128 | 123 | 140
  Week 5 | -12.0 (9.24) | -11.9 (9.69) | -14.9 (8.91)
  Week 6: number analyzed (Participants) | 129 | 116 | 136
  Week 6 | -14.3 (9.98) | -14.5 (10.59) | -17.3 (8.75)
  Week 8: number analyzed (Participants) | 116 | 103 | 133
  Week 8 | -15.1 (10.09) | -17.3 (9.65) | -19.1 (9.14)

16. Secondary Outcome: Mean Change From Randomization in IDS-CR Total Score Over Week 8
Description: The IDS-CR is a standardized 30-item, clinician rated scale to assess the severity of a participant's depressive symptoms. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. In order to calculate the total score of IDS-CR, the following procedures were used: either item 11 or 12 were scored; either item 13 or 14 were scored; if both items 11 and 12 (or 13 and 14) were scored, the highest of the items was scored. The total score was obtained by adding the scores of 28 items of the 30 items. Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between IDS-CR total score at the time points being analyzed (Week 1, 2, 3, 4, 5, 6 and 8) to Randomization.
Time Frame: Week 0 (Randomization) up to Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 150 | 167 | 164
  Week 1 | -4.4 (7.16) | -4.9 (7.54) | -5.1 (8.56)
  Week 2: number analyzed (Participants) | 145 | 151 | 152
  Week 2 | -8.8 (9.03) | -9.7 (10.37) | -9.8 (11.55)
  Week 3: number analyzed (Participants) | 137 | 144 | 151
  Week 3 | -12.7 (11.07) | -11.2 (11.36) | -14.3 (11.90)
  Week 4: number analyzed (Participants) | 138 | 138 | 147
  Week 4 | -15.0 (12.42) | -13.2 (10.97) | -16.2 (11.80)
  Week 5: number analyzed (Participants) | 128 | 123 | 140
  Week 5 | -16.9 (11.51) | -16.9 (13.07) | -20.1 (12.05)
  Week 6: number analyzed (Participants) | 129 | 116 | 136
  Week 6 | -19.5 (13.11) | -19.3 (14.40) | -23.4 (12.60)
  Week 8: number analyzed (Participants) | 116 | 103 | 133
  Week 8 | -20.3 (14.81) | -22.8 (14.09) | -25.2 (12.77)

17. Secondary Outcome: Mean Change From Randomization in the in Bech Scale (6-item of HAMD-17 Scale) Score Over Week 8
Description: The HAMD is a rating instrument for evaluating severity of symptoms of depression, was completed by the participant. Rating instrument used in this study was the 17-item version (HAM-D17). The Bech scale of the HAMD-17 is composed of 6 identified items out of the 17 items rated in HAMD-17 scale. Each item is rated on either a 3-point scale (0 to 2) or a 5-point scale (0 to 4). The following symptoms were rated on a 5-point scale (0-4): depressed mood, feeling of guilt, work and interests, psychomotor retardation, and anxiety (psychic). The following symptom was rated on a 3-point scale (0-2): somatic symptoms (general). Total score ranged from 0 to 22, with 0 indicating absence of symptoms and a higher score indicating greater severity of symptoms. Randomization value was defined as the assessment value done on Week 0. Change from Randomization in total score was the difference between Bech total score at the time points being analyzed (Week 1, 2, 3, 4, 5, 6 and 8) to randomization.
Time Frame: Week 0 (Randomization) up to Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Score on scale
  Week 1: number analyzed (Participants) | 150 | 167 | 164
  Week 1 | -0.8 (2.06) | -1.0 (2.55) | -1.2 (2.52)
  Week 2: number analyzed (Participants) | 145 | 151 | 152
  Week 2 | -2.0 (2.58) | -2.2 (3.25) | -2.6 (3.28)
  Week 3: number analyzed (Participants) | 137 | 144 | 151
  Week 3 | -3.3 (3.10) | -2.8 (3.82) | -3.8 (3.56)
  Week 4: number analyzed (Participants) | 138 | 138 | 147
  Week 4 | -3.9 (3.62) | -3.5 (3.60) | -4.3 (3.63)
  Week 5: number analyzed (Participants) | 128 | 123 | 140
  Week 5 | -4.4 (3.42) | -4.4 (4.26) | -5.6 (3.61)
  Week 6: number analyzed (Participants) | 128 | 116 | 136
  Week 6 | -5.1 (4.03) | -5.4 (4.44) | -6.5 (3.78)
  Week 8 | -5.3 (4.19) | -6.3 (4.10) | -7.2 (3.92)

18. Secondary Outcome: Percentage of Responders and Remitters of MADRS Over Week 10
Description: The MADRS scale measures the depression level of a participant. The total score was derived by adding the scores of the following 10 items: 1, apparent sadness; 2, reported sadness; 3, inner tension; 4, reduced sleep; 5, reduced appetite; 6, concentration difficulties; 7, lassitude; 8, inability to feel; 9, pessimistic thoughts; 10, suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). The total score ranged from 0-60, where 0 indicated no depression and 60 indicated severely depressed. Responders were defined as participants who had a >=50% reduction from randomization in MADRS total Score. Percentage change from randomization was calculated as total score at post Randomization visit minus total score at Randomization visit divided by total score at Randomization visit multiplied by 100. Remitters were defined as participants with a MADRS total score <=11.
Time Frame: Up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Percentage of participants
  Responders, Week 1: number analyzed (Participants) | 150 | 167 | 164
  Responders, Week 1 | 3 | 3 | 4
  Responders, Week 2: number analyzed (Participants) | 145 | 151 | 152
  Responders, Week 2 | 8 | 11 | 13
  Responders, Week 3: number analyzed (Participants) | 137 | 144 | 151
  Responders, Week 3 | 20 | 14 | 25
  Responders, Week 4: number analyzed (Participants) | 138 | 138 | 147
  Responders, Week 4 | 29 | 17 | 35
  Responders, Week 5: number analyzed (Participants) | 128 | 123 | 140
  Responders, Week 5 | 35 | 35 | 51
  Responders, Week 6: number analyzed (Participants) | 129 | 116 | 136
  Responders, Week 6 | 40 | 41 | 63
  Responders, Week 8: number analyzed (Participants) | 116 | 103 | 133
  Responders, Week 8 | 44 | 54 | 72
  Responders, Week 10: number analyzed (Participants) | 117 | 100 | 130
  Responders, Week 10 | 55 | 64 | 81
  Remitters, Week 1: number analyzed (Participants) | 150 | 167 | 164
  Remitters, Week 1 | 2 | 3 | 3
  Remitters, Week 2: number analyzed (Participants) | 145 | 151 | 152
  Remitters, Week 2 | 5 | 7 | 11
  Remitters, Week 3: number analyzed (Participants) | 137 | 144 | 151
  Remitters, Week 3 | 12 | 10 | 17
  Remitters, Week 4: number analyzed (Participants) | 138 | 138 | 147
  Remitters, Week 4 | 18 | 12 | 22
  Remitters, Week 5: number analyzed (Participants) | 128 | 123 | 140
  Remitters, Week 5 | 17 | 24 | 38
  Remitters, Week 6: number analyzed (Participants) | 129 | 116 | 136
  Remitters, Week 6 | 28 | 33 | 48
  Remitters, Week 8: number analyzed (Participants) | 116 | 103 | 133
  Remitters, Week 8 | 35 | 41 | 55
  Remitters, Week 10: number analyzed (Participants) | 117 | 100 | 130
  Remitters, Week 10 | 45 | 52 | 68
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS responders at Week 1; Test type: Superiority or Other; p = 0.5061, Generalized estimating equation model; Odds Ratio (OR) = 0.64, 90% CI 2-sided [0.21 to 1.93]
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS responders at Week 1; Test type: Superiority or Other; p = 0.7398, Generalized estimating equation model; Odds Ratio (OR) = 1.22, 90% CI 2-sided [0.46 to 3.25]
Statistical Analysis 3: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS responders at Week 2; Test type: Superiority or Other; p = 0.9209, Generalized estimating equation model; Odds Ratio (OR) = 1.04, 90% CI 2-sided [0.52 to 2.08]
Statistical Analysis 4: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS responders at Week 2; Test type: Superiority or Other; p = 0.2908, Generalized estimating equation model; Odds Ratio (OR) = 1.56, 90% CI 2-sided [0.78 to 3.13]
Statistical Analysis 5: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS responders at Week 3; Test type: Superiority or Other; p = 0.0086, Generalized estimating equation model; Odds Ratio (OR) = 0.41, 90% CI 2-sided [0.23 to 0.72]
Statistical Analysis 6: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS responders at Week 3; Test type: Superiority or Other; p = 0.8087, Generalized estimating equation model; Odds Ratio (OR) = 1.08, 90% CI 2-sided [0.64 to 1.83]
Statistical Analysis 7: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS responders at Week 4; Test type: Superiority or Other; p = 0.0002, Generalized estimating equation model; Odds Ratio (OR) = 0.31, 90% CI 2-sided [0.18 to 0.52]
Statistical Analysis 8: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS responders at Week 4; Test type: Superiority or Other; p = 0.4606, Generalized estimating equation model; Odds Ratio (OR) = 1.23, 90% CI 2-sided [0.78 to 1.94]
Statistical Analysis 9: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS responders at Week 5; Test type: Superiority or Other; p = 0.1399, Generalized estimating equation model; Odds Ratio (OR) = 0.65, 90% CI 2-sided [0.40 to 1.05]
Statistical Analysis 10: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS responders at Week 5; Test type: Superiority or Other; p = 0.0461, Generalized estimating equation model; Odds Ratio (OR) = 1.73, 90% CI 2-sided [1.10 to 2.73]
Statistical Analysis 11: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS responders at Week 6; Test type: Superiority or Other; p = 0.1400, Generalized estimating equation model; Odds Ratio (OR) = 0.66, 90% CI 2-sided [0.41 to 1.05]
Statistical Analysis 12: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS responders at Week 6; Test type: Superiority or Other; p = 0.0002, Generalized estimating equation model; Odds Ratio (OR) = 2.71, 90% CI 2-sided [1.74 to 4.21]
Statistical Analysis 13: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS responders at Week 8; Test type: Superiority or Other; p = 0.9596, Generalized estimating equation model; Odds Ratio (OR) = 0.98, 90% CI 2-sided [0.59 to 1.64]
Statistical Analysis 14: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS responders at Week 8; Test type: Superiority or Other; p = 0.0000, Generalized estimating equation model; Odds Ratio (OR) = 3.24, 90% CI 2-sided [2.01 to 5.23]
Statistical Analysis 15: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS responders at Week 10; Test type: Superiority or Other; p = 0.6530, Generalized estimating equation model; Odds Ratio (OR) = 1.15, 90% CI 2-sided [0.69 to 1.93]
Statistical Analysis 16: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS responders at Week 10; Test type: Superiority or Other; p = 0.0000, Generalized estimating equation model; Odds Ratio (OR) = 3.48, 90% CI 2-sided [2.11 to 5.73]
Statistical Analysis 17: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS remitters at Week 1; Test type: Superiority or Other; p = 0.8844, Generalized estimating equation model; Odds Ratio (OR) = 0.89, 90% CI 2-sided [0.23 to 3.48]
Statistical Analysis 18: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS remitters at Week 1; Test type: Superiority or Other; p = 0.7425, Generalized estimating equation model; Odds Ratio (OR) = 1.29, 90% CI 2-sided [0.36 to 4.68]
Statistical Analysis 19: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS remitters at Week 2; Test type: Superiority or Other; p = 0.8355, Generalized estimating equation model; Odds Ratio (OR) = 0.90, 90% CI 2-sided [0.39 to 2.07]
Statistical Analysis 20: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS remitters at Week 2; Test type: Superiority or Other; p = 0.1786, Generalized estimating equation model; Odds Ratio (OR) = 1.93, 90% CI 2-sided [0.86 to 4.32]
Statistical Analysis 21: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS remitters at Week 3; Test type: Superiority or Other; p = 0.0835, Generalized estimating equation model; Odds Ratio (OR) = 0.50, 90% CI 2-sided [0.26 to 0.97]
Statistical Analysis 22: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS remitters at Week 3; Test type: Superiority or Other; p = 0.8558, Generalized estimating equation model; Odds Ratio (OR) = 1.07, 90% CI 2-sided [0.58 to 1.98]
Statistical Analysis 23: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS remitters at Week 4; Test type: Superiority or Other; p = 0.0067, Generalized estimating equation model; Odds Ratio (OR) = 0.36, 90% CI 2-sided [0.20 to 0.67]
Statistical Analysis 24: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS remitters at Week 4; Test type: Superiority or Other; p = 0.6647, Generalized estimating equation model; Odds Ratio (OR) = 1.15, 90% CI 2-sided [0.67 to 1.98]
Statistical Analysis 25: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS remitters at Week 5; Test type: Superiority or Other; p = 0.9553, Generalized estimating equation model; Odds Ratio (OR) = 0.98, 90% CI 2-sided [0.55 to 1.74]
Statistical Analysis 26: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS remitters at Week 5; Test type: Superiority or Other; p = 0.0040, Generalized estimating equation model; Odds Ratio (OR) = 2.58, 90% CI [1.50 to 4.42]
Statistical Analysis 27: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS remitters at Week 6; Test type: Superiority or Other; p = 0.6327, Generalized estimating equation model; Odds Ratio (OR) = 0.86, 90% CI 2-sided [0.52 to 1.43]
Statistical Analysis 28: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS remitters at Week 6; Test type: Superiority or Other; p = 0.0027, Generalized estimating equation model; Odds Ratio (OR) = 2.36, 90% CI 2-sided [1.47 to 3.79]
Statistical Analysis 29: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS remitters at Week 8; Test type: Superiority or Other; p = 0.3961, Generalized estimating equation model; Odds Ratio (OR) = 0.76, 90% CI 2-sided [0.45 to 1.29]
Statistical Analysis 30: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS remitters at Week 8; Test type: Superiority or Other; p = 0.0298, Generalized estimating equation model; Odds Ratio (OR) = 1.89, 90% CI 2-sided [1.17 to 3.06]
Statistical Analysis 31: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in MADRS remitters at Week 10; Test type: Superiority or Other; p = 0.8826, Generalized estimating equation model; Odds Ratio (OR) = 0.95, 90% CI 2-sided [0.56 to 1.61]
Statistical Analysis 32: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in MADRS remitters at Week 10; Test type: Superiority or Other; p = 0.0022, Generalized estimating equation model; Odds Ratio (OR) = 2.48, 90% CI 2-sided [1.52 to 4.05]

19. Secondary Outcome: Percentage of Responders and Remitters of IDS-CR Over Week 10
Description: IDS-CR is a standardized 30-item, clinician rated scale to assess the severity of a participant's depressive symptoms. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Total score of IDS-CR calculated as : either item 11 or 12 scored; either item 13 or 14 scored; if both items scored, the highest of the items was used. Total score was obtained by adding the scores of 28 items of the 30 items. Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression. Responders were defined as participants who had a >=50% reduction from randomization in IDS-CR total Score. Percentage change from randomization was calculated as total score at post Randomization visit minus total score at Randomization visit divided by total score at Randomization visit multiplied by 100. Remitters were defined as participants with a IDS-CR total score <=14.
Time Frame: Up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Percentage of participants
  Responders, Week 1: number analyzed (Participants) | 150 | 167 | 164
  Responders, Week 1 | 4 | 3 | 5
  Responders, Week 2: number analyzed (Participants) | 145 | 151 | 152
  Responders, Week 2 | 8 | 11 | 14
  Responders, Week 3: number analyzed (Participants) | 137 | 144 | 151
  Responders, Week 3 | 17 | 15 | 26
  Responders, Week 4: number analyzed (Participants) | 138 | 138 | 147
  Responders, Week 4 | 25 | 17 | 33
  Responders, Week 5: number analyzed (Participants) | 128 | 123 | 140
  Responders, Week 5 | 28 | 31 | 44
  Responders, Week 6: number analyzed (Participants) | 129 | 116 | 136
  Responders, Week 6 | 36 | 37 | 58
  Responders, Week 8: number analyzed (Participants) | 116 | 103 | 133
  Responders, Week 8 | 43 | 50 | 62
  Responders, Week 10: number analyzed (Participants) | 117 | 100 | 130
  Responders, Week 10 | 50 | 60 | 72
  Remitters, Week 1: number analyzed (Participants) | 150 | 167 | 164
  Remitters, Week 1 | 3 | 1 | 1
  Remitters, Week 2: number analyzed (Participants) | 145 | 151 | 152
  Remitters, Week 2 | 3 | 8 | 8
  Remitters, Week 3: number analyzed (Participants) | 137 | 144 | 151
  Remitters, Week 3 | 8 | 8 | 13
  Remitters, Week 4: number analyzed (Participants) | 138 | 138 | 147
  Remitters, Week 4 | 17 | 10 | 16
  Remitters, Week 5: number analyzed (Participants) | 128 | 123 | 140
  Remitters, Week 5 | 16 | 18 | 27
  Remitters, Week 6: number analyzed (Participants) | 129 | 116 | 136
  Remitters, Week 6 | 22 | 21 | 40
  Remitters, Week 8: number analyzed (Participants) | 116 | 103 | 133
  Remitters, Week 8 | 28 | 31 | 44
  Remitters, Week 10: number analyzed (Participants) | 117 | 100 | 130
  Remitters, Week 10 | 35 | 38 | 48
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR responders at Week 1; Test type: Superiority or Other; p = 0.5072, Generalized estimating equation model; Odds Ratio (OR) = 0.65, 90% CI 2-sided [0.22 to 1.89]
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR responders at Week 1; Test type: Superiority or Other; p = 0.6886, Generalized estimating equation model; Odds Ratio (OR) = 1.23, 90% CI 2-sided [0.52 to 2.93]
Statistical Analysis 3: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR responders at Week 2; Test type: Superiority or Other; p = 0.8664, Generalized estimating equation model; Odds Ratio (OR) = 1.07, 90% CI 2-sided [0.56 to 2.04]
Statistical Analysis 4: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR responders at Week 2; Test type: Superiority or Other; p = 0.2897, Generalized estimating equation model; Odds Ratio (OR) = 1.50, 90% CI 2-sided [0.80 to 2.79]
Statistical Analysis 5: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR responders at Week 3; Test type: Superiority or Other; p = 0.2474, Generalized estimating equation model; Odds Ratio (OR) = 0.68, 90% CI 2-sided [0.39 to 1.18]
Statistical Analysis 6: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR responders at Week 3; Test type: Superiority or Other; p = 0.2007, Generalized estimating equation model; Odds Ratio (OR) = 1.49, 90% CI 2-sided [0.89 to 2.47]
Statistical Analysis 7: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR responders at Week 4; Test type: Superiority or Other; p = 0.0214, Generalized estimating equation model; Odds Ratio (OR) = 0.49, 90% CI 2-sided [0.29 to 0.82]
Statistical Analysis 8: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR responders at Week 4; Test type: Superiority or Other; p = 0.2368, Generalized estimating equation model; Odds Ratio (OR) = 1.40, 90% CI 2-sided [0.88 to 2.23]
Statistical Analysis 9: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR responders at Week 5; Test type: Superiority or Other; p = 0.9870, Generalized estimating equation model; Odds Ratio (OR) = 1.00, 90% CI 2-sided [0.63 to 1.59]
Statistical Analysis 10: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR responders at Week 5; Test type: Superiority or Other; p = 0.0193, Generalized estimating equation model; Odds Ratio (OR) = 1.91, 90% CI 2-sided [1.21 to 3.00]
Statistical Analysis 11: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR responders at Week 6; Test type: Superiority or Other; p = 0.8351, Generalized estimating equation model; Odds Ratio (OR) = 0.94, 90% CI 2-sided [0.59 to 1.50]
Statistical Analysis 12: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR responders at Week 6; Test type: Superiority or Other; p = 0.0001, Generalized estimating equation model; Odds Ratio (OR) = 3.01, 90% CI 2-sided [1.90 to 4.77]
Statistical Analysis 13: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR responders at Week 8; Test type: Superiority or Other; p = 0.7510, Generalized estimating equation model; Odds Ratio (OR) = 1.10, 90% CI 2-sided [0.67 to 1.80]
Statistical Analysis 14: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR responders at Week 8; Test type: Superiority or Other; p = 0.0029, Generalized estimating equation model; Odds Ratio (OR) = 2.37, 90% CI 2-sided [1.47 to 3.80]
Statistical Analysis 15: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR responders at Week 10; Test type: Superiority or Other; p = 0.1707, Generalized estimating equation model; Odds Ratio (OR) = 1.53, 90% CI 2-sided [0.92 to 2.55]
Statistical Analysis 16: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR responders at Week 10; Test type: Superiority or Other; p = 0.0001, Generalized estimating equation model; Odds Ratio (OR) = 3.27, 90% CI 2-sided [1.99 to 5.36]
Statistical Analysis 17: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR remitters at Week 1; Test type: Superiority or Other; p = 0.2050, Generalized estimating equation model; Odds Ratio (OR) = 0.27, 90% CI 2-sided [0.05 to 1.48]
Statistical Analysis 18: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR remitters at Week 1; Test type: Superiority or Other; p = 0.1735, Generalized estimating equation model; Odds Ratio (OR) = 0.36, 90% CI 2-sided [0.11 to 1.24]
Statistical Analysis 19: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR remitters at Week 2; Test type: Superiority or Other; p = 0.2305, Generalized estimating equation model; Odds Ratio (OR) = 1.93, 90% CI 2-sided [0.78 to 4.75]
Statistical Analysis 20: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR remitters at Week 2; Test type: Superiority or Other; p = 0.2507, Generalized estimating equation model; Odds Ratio (OR) = 1.86, 90% CI 2-sided [0.77 to 4.50]
Statistical Analysis 21: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR remitters at Week 3; Test type: Superiority or Other; p = 0.5608, Generalized estimating equation model; Odds Ratio (OR) = 0.76, 90% CI 2-sided [0.35 to 1.64]
Statistical Analysis 22: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR remitters at Week 3; Test type: Superiority or Other; p = 0.6526, Generalized estimating equation model; Odds Ratio (OR) = 1.21, 90% CI 2-sided [0.60 to 2.42]
Statistical Analysis 23: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR remitters at Week 4; Test type: Superiority or Other; p = 0.0208, Generalized estimating equation model; Odds Ratio (OR) = 0.41, 90% CI 2-sided [0.21 to 0.77]
Statistical Analysis 24: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR remitters at Week 4; Test type: Superiority or Other; p = 0.2859, Generalized estimating equation model; Odds Ratio (OR) = 0.69, 90% CI 2-sided [0.39 to 1.22]
Statistical Analysis 25: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR remitters at Week 5; Test type: Superiority or Other; p = 0.7921, Generalized estimating equation model; Odds Ratio (OR) = 0.91, 90% CI 2-sided [0.49 to 1.66]
Statistical Analysis 26: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR remitters at Week 5; Test type: Superiority or Other; p = 0.3620, Generalized estimating equation model; Odds Ratio (OR) = 1.35, 90% CI 2-sided [0.79 to 2.31]
Statistical Analysis 27: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR remitters at Week 6; Test type: Superiority or Other; p = 0.4331, Generalized estimating equation model; Odds Ratio (OR) = 0.77, 90% CI 2-sided [0.44 to 1.34]
Statistical Analysis 28: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR remitters at Week 6; Test type: Superiority or Other; p = 0.0047, Generalized estimating equation model; Odds Ratio (OR) = 2.30, 90% CI 2-sided [1.42 to 3.75]
Statistical Analysis 29: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR remitters at Week 8; Test type: Superiority or Other; p = 0.4431, Generalized estimating equation model; Odds Ratio (OR) = 0.78, 90% CI 2-sided [0.46 to 1.32]
Statistical Analysis 30: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR remitters at Week 8; Test type: Superiority or Other; p = 0.1901, Generalized estimating equation model; Odds Ratio (OR) = 1.48, 90% CI 2-sided [0.90 to 2.44]
Statistical Analysis 31: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in IDS-CR remitters at Week 10; Test type: Superiority or Other; p = 0.9222, Generalized estimating equation model; Odds Ratio (OR) = 0.97, 90% CI 2-sided [0.56 to 1.66]
Statistical Analysis 32: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in IDS-CR remitters at Week 10; Test type: Superiority or Other; p = 0.1665, Generalized estimating equation model; Odds Ratio (OR) = 1.50, 90% CI 2-sided [0.93 to 2.43]

20. Secondary Outcome: Percentage of Responders and Remitters of HAMD-17 Over Week 10
Description: HAMD-17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, work and activities, sleep, suicide, psychomotor agitation/retardation, appetite, sexual interest, anxiety, and somatic symptoms). The items of the HAMD-17 are rated on a scale of 0 to 2 or 0 to 4, and the total score ranges from 0 to 52, where 0 indicates absence of symptom and higher scores indicates more severe symptoms. Responders were defined as participants who had a >=50% reduction from randomization in HAMD-17 total Score. Percentage change from randomization was calculated as total score at post Randomization visit minus total score at Randomization visit divided by total score at Randomization visit multiplied by 100. Remitters were defined as participants with a HAMD-17 total score <=7.
Time Frame: Up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Percentage of participants
  Responders, Week 1: number analyzed (Participants) | 150 | 167 | 164
  Responders, Week 1 | 3 | 2 | 4
  Responders, Week 2: number analyzed (Participants) | 145 | 151 | 152
  Responders, Week 2 | 8 | 10 | 14
  Responders, Week 3: number analyzed (Participants) | 137 | 144 | 151
  Responders, Week 3 | 16 | 14 | 25
  Responders, Week 4: number analyzed (Participants) | 138 | 138 | 147
  Responders, Week 4 | 25 | 14 | 32
  Responders, Week 5: number analyzed (Participants) | 128 | 123 | 140
  Responders, Week 5 | 29 | 30 | 42
  Responders, Week 6: number analyzed (Participants) | 129 | 116 | 136
  Responders, Week 6 | 36 | 33 | 54
  Responders, Week 8: number analyzed (Participants) | 116 | 103 | 133
  Responders, Week 8 | 41 | 48 | 62
  Responders, Week 10: number analyzed (Participants) | 117 | 100 | 130
  Responders, Week 10 | 51 | 55 | 72
  Remitters, Week 1: number analyzed (Participants) | 150 | 167 | 164
  Remitters, Week 1 | 2 | 2 | 2
  Remitters, Week 2: number analyzed (Participants) | 145 | 151 | 152
  Remitters, Week 2 | 3 | 5 | 9
  Remitters, Week 3: number analyzed (Participants) | 137 | 144 | 151
  Remitters, Week 3 | 7 | 8 | 15
  Remitters, Week 4: number analyzed (Participants) | 138 | 138 | 147
  Remitters, Week 4 | 17 | 9 | 16
  Remitters, Week 5: number analyzed (Participants) | 128 | 123 | 140
  Remitters, Week 5 | 16 | 15 | 26
  Remitters, Week 6: number analyzed (Participants) | 129 | 116 | 136
  Remitters, Week 6 | 23 | 20 | 40
  Remitters, Week 8: number analyzed (Participants) | 116 | 103 | 133
  Remitters, Week 8 | 28 | 29 | 45
  Remitters, Week 10: number analyzed (Participants) | 117 | 100 | 130
  Remitters, Week 10 | 35 | 39 | 52
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 responders at Week 1; Test type: Superiority or Other; p = 0.5057, Generalized estimating equation model; Odds Ratio (OR) = 0.63, 90% CI 2-sided [0.20 to 1.98]
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 responders at Week 1; Test type: Superiority or Other; p = 0.8633, Generalized estimating equation model; Odds Ratio (OR) = 1.12, 90% CI 2-sided [0.38 to 3.30]
Statistical Analysis 3: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 responders at Week 2; Test type: Superiority or Other; p = 0.8428, Generalized estimating equation model; Odds Ratio (OR) = 1.09, 90% CI 2-sided [0.55 to 2.16]
Statistical Analysis 4: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 responders at Week 2; Test type: Superiority or Other; p = 0.3416, Generalized estimating equation model; Odds Ratio (OR) = 1.47, 90% CI 2-sided [0.76 to 2.84]
Statistical Analysis 5: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 responders at Week 3; Test type: Superiority or Other; p = 0.3287, Generalized estimating equation model; Odds Ratio (OR) = 0.71, 90% CI 2-sided [0.40 to 1.26]
Statistical Analysis 6: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 responders at Week 3; Test type: Superiority or Other; p = 0.2112, Generalized estimating equation model; Odds Ratio (OR) = 1.50, 90% CI 2-sided [0.88 to 2.57]
Statistical Analysis 7: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 responders at Week 4; Test type: Superiority or Other; p = 0.0134, Generalized estimating equation model; Odds Ratio (OR) = 0.44, 90% CI 2-sided [0.26 to 0.76]
Statistical Analysis 8: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 responders at Week 4; Test type: Superiority or Other; p = 0.3412, Generalized estimating equation model; Odds Ratio (OR) = 1.33, 90% CI 2-sided [0.81 to 2.17]
Statistical Analysis 9: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 responders at Week 5; Test type: Superiority or Other; p = 0.8434, Generalized estimating equation model; Odds Ratio (OR) = 0.94, 90% CI 2-sided [0.58 to 1.54]
Statistical Analysis 10: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 responders at Week 5; Test type: Superiority or Other; p = 0.0819, Generalized estimating equation model; Odds Ratio (OR) = 1.65, 90% CI 2-sided [1.03 to 2.63]
Statistical Analysis 11: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 responders at Week 6; Test type: Superiority or Other; p = 0.2832, Generalized estimating equation model; Odds Ratio (OR) = 0.72, 90% CI 2-sided [0.44 to 1.19]
Statistical Analysis 12: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 responders at Week 6; Test type: Superiority or Other; p = 0.0016, Generalized estimating equation model; Odds Ratio (OR) = 2.47, 90% CI 2-sided [1.54 to 3.97]
Statistical Analysis 13: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 responders at Week 8; Test type: Superiority or Other; p = 0.9727, Generalized estimating equation model; Odds Ratio (OR) = 0.99, 90% CI 2-sided [0.60 to 1.63]
Statistical Analysis 14: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 responders at Week 8; Test type: Superiority or Other; p = 0.0010, Generalized estimating equation model; Odds Ratio (OR) = 2.57, 90% CI 2-sided [1.60 to 4.13]
Statistical Analysis 15: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 responders at Week 10; Test type: Superiority or Other; p = 0.8312, Generalized estimating equation model; Odds Ratio (OR) = 1.07, 90% CI 2-sided [0.64 to 1.80]
Statistical Analysis 16: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 responders at Week 10; Test type: Superiority or Other; p = 0.0002, Generalized estimating equation model; Odds Ratio (OR) = 3.06, 90% CI 2-sided [1.86 to 5.02]
Statistical Analysis 17: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 remitters at Week 1; Test type: Superiority or Other; p = 0.5530, Generalized estimating equation model; Odds Ratio (OR) = 0.58, 90% CI 2-sided [0.13 to 2.60]
Statistical Analysis 18: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 remitters at Week 1; Test type: Superiority or Other; p = 0.9780, Generalized estimating equation model; Odds Ratio (OR) = 0.98, 90% CI 2-sided [0.28 to 3.41]
Statistical Analysis 19: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 remitters at Week 2; Test type: Superiority or Other; p = 0.8312, Generalized estimating equation model; Odds Ratio (OR) = 1.14, 90% CI 2-sided [0.43 to 3.03]
Statistical Analysis 20: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 remitters at Week 2; Test type: Superiority or Other; p = 0.1881, Generalized estimating equation model; Odds Ratio (OR) = 2.09, 90% CI 2-sided [0.83 to 5.25]
Statistical Analysis 21: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 remitters at Week 3; Test type: Superiority or Other; p = 0.6384, Generalized estimating equation model; Odds Ratio (OR) = 0.81, 90% CI 2-sided [0.39 to 1.69]
Statistical Analysis 22: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 remitters at Week 3; Test type: Superiority or Other; p = 0.2160, Generalized estimating equation model; Odds Ratio (OR) = 1.68, 90% CI 2-sided [0.84 to 3.37]
Statistical Analysis 23: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 remitters at Week 4; Test type: Superiority or Other; p = 0.0259, Generalized estimating equation model; Odds Ratio (OR) = 0.40, 90% CI 2-sided [0.20 to 0.79]
Statistical Analysis 24: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 remitters at Week 4; Test type: Superiority or Other; p = 0.3959, Generalized estimating equation model; Odds Ratio (OR) = 0.73, 90% CI 2-sided [0.39 to 1.35]
Statistical Analysis 25: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 remitters at Week 5; Test type: Superiority or Other; p = 0.3857, Generalized estimating equation model; Odds Ratio (OR) = 0.72, 90% CI 2-sided [0.39 to 1.34]
Statistical Analysis 26: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 remitters at Week 5; Test type: Superiority or Other; p = 0.3126, Generalized estimating equation model; Odds Ratio (OR) = 1.42, 90% CI 2-sided [0.80 to 2.52]
Statistical Analysis 27: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 remitters at Week 6; Test type: Superiority or Other; p = 0.1182, Generalized estimating equation model; Odds Ratio (OR) = 0.61, 90% CI 2-sided [0.36 to 1.03]
Statistical Analysis 28: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 remitters at Week 6; Test type: Superiority or Other; p = 0.0125, Generalized estimating equation model; Odds Ratio (OR) = 2.10, 90% CI 2-sided [1.29 to 3.43]
Statistical Analysis 29: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 remitters at Week 8; Test type: Superiority or Other; p = 0.2147, Generalized estimating equation model; Odds Ratio (OR) = 0.69, 90% CI 2-sided [0.42 to 1.13]
Statistical Analysis 30: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 remitters at Week 8; Test type: Superiority or Other; p = 0.0783, Generalized estimating equation model; Odds Ratio (OR) = 1.67, 90% CI 2-sided [1.03 to 2.69]
Statistical Analysis 31: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in HAMD-17 remitters at Week 10; Test type: Superiority or Other; p = 0.9067, Generalized estimating equation model; Odds Ratio (OR) = 0.96, 90% CI [0.57 to 1.64]
Statistical Analysis 32: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in HAMD-17 remitters at Week 10; Test type: Superiority or Other; p = 0.0328, Generalized estimating equation model; Odds Ratio (OR) = 1.83, 90% CI 2-sided [1.15 to 2.92]

21. Secondary Outcome: Percentage of Participants With Clinical Global Impression - Global Improvement (CGI-I) Over Week 10
Description: The CGI-I scale measures the improvement of psychiatric symptoms on a 7-point scale from 1-7. The scale was rated by the clinician at every visit during the treatment phase (Week 1 through Week 10/early withdrawal) of the participant's total improvement or worsening compared with that individual's condition at the start of the study (the Randomization visit , Week 0) whether or not the change is judged to be due to drug treatment. The scores indicated the following: 1= very much improved; 2= much improved; 3= minimally improved; 4= no change; 5= minimally worse; 6= much worse; 7= very much worse. The score ranged from 1-7, where 1 indicated very much improved and higher score indicated greater severity of symptoms. Randomization value was defined as the assessment value done on Week 0. Data is reported for the percentage of participants who were much improved and very much improved.
Time Frame: Up to Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Percentage of participants
  Week 1: number analyzed (Participants) | 150 | 168 | 164
  Week 1 | 3 | 4 | 5
  Week 2: number analyzed (Participants) | 145 | 151 | 153
  Week 2 | 12 | 17 | 20
  Week 3: number analyzed (Participants) | 138 | 145 | 152
  Week 3 | 28 | 27 | 41
  Week 4: number analyzed (Participants) | 138 | 138 | 147
  Week 4 | 40 | 36 | 49
  Week 5: number analyzed (Participants) | 128 | 123 | 140
  Week 5 | 45 | 48 | 66
  Week 6: number analyzed (Participants) | 129 | 117 | 136
  Week 6 | 59 | 59 | 77
  Week 8: number analyzed (Participants) | 117 | 105 | 133
  Week 8 | 61 | 69 | 83
  Week 10: number analyzed (Participants) | 117 | 100 | 130
  Week 10 | 62 | 75 | 82
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in percentage of participants with CGI-I at Week 1; Test type: Superiority or Other; p = 0.6928, Generalized estimating equation model; Odds Ratio (OR) = 1.29, 90% CI 2-sided [0.44 to 3.76]
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in percentage of participants with CGI-I at Week 1; Test type: Superiority or Other; p = 0.3039, Generalized estimating equation model; Odds Ratio (OR) = 1.86, 90% CI 2-sided [0.69 to 5.01]
Statistical Analysis 3: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in percentage of participants with CGI-I at Week 2; Test type: Superiority or Other; p = 0.1938, Generalized estimating equation model; Odds Ratio (OR) = 1.55, 90% CI 2-sided [0.89 to 2.70]
Statistical Analysis 4: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in percentage of participants with CGI-I at Week 2; Test type: Superiority or Other; p = 0.0600, Generalized estimating equation model; Odds Ratio (OR) = 1.85, 90% CI 2-sided [1.08 to 3.16]
Statistical Analysis 5: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in percentage of participants with CGI-I at Week 3; Test type: Superiority or Other; p = 0.8989, Generalized estimating equation model; Odds Ratio (OR) = 0.96, 90% CI 2-sided [0.61 to 1.53]
Statistical Analysis 6: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in percentage of participants with CGI-I at Week 3; Test type: Superiority or Other; p = 0.0136, Generalized estimating equation model; Odds Ratio (OR) = 1.95, 90% CI 2-sided [1.25 to 3.05]
Statistical Analysis 7: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in percentage of participants with CGI-I at Week 4; Test type: Superiority or Other; p = 0.3099, Generalized estimating equation model; Odds Ratio (OR) = 0.77, 90% CI 2-sided [0.50 to 1.18]
Statistical Analysis 8: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in percentage of participants with CGI-I at Week 4; Test type: Superiority or Other; p = 0.1137, Generalized estimating equation model; Odds Ratio (OR) = 1.49, 90% CI 2-sided [0.98 to 2.27]
Statistical Analysis 9: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in percentage of participants with CGI-I at Week 5; Test type: Superiority or Other; p = 0.8682, Generalized estimating equation model; Odds Ratio (OR) = 1.05, 90% CI [0.67 to 1.64]
Statistical Analysis 10: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in percentage of participants with CGI-I at Week 5; Test type: Superiority or Other; p = 0.0006, Generalized estimating equation model; Odds Ratio (OR) = 2.56, 90% CI 2-sided [1.63 to 4.03]
Statistical Analysis 11: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in percentage of participants with CGI-I at Week 6; Test type: Superiority or Other; p = 0.8992, Generalized estimating equation model; Odds Ratio (OR) = 0.97, 90% CI 2-sided [0.62 to 1.51]
Statistical Analysis 12: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in percentage of participants with CGI-I at Week 6; Test type: Superiority or Other; p = 0.0004, Generalized estimating equation model; Odds Ratio (OR) = 2.61, 90% CI 2-sided [1.67 to 4.09]
Statistical Analysis 13: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in percentage of participants with CGI-I at Week 8; Test type: Superiority or Other; p = 0.2800, Placebo versus GSK372475 in percentage o; Odds Ratio (OR) = 1.37, 90% CI 2-sided [0.85 to 2.23]
Statistical Analysis 14: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in percentage of participants with CGI-I at Week 8; Test type: Superiority or Other; p = 0.0000, Generalized estimating equation model; Odds Ratio (OR) = 3.69, 90% CI 2-sided [2.24 to 6.08]
Statistical Analysis 15: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in percentage of participants with CGI-I at Week 10; Test type: Superiority or Other; p = 0.0507, Generalized estimating equation model; Odds Ratio (OR) = 1.86, 90% CI 2-sided [1.10 to 3.13]
Statistical Analysis 16: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in percentage of participants with CGI-I at Week 10; Test type: Superiority or Other; p = 0.0003, Generalized estimating equation model; Odds Ratio (OR) = 2.97, 90% CI 2-sided [1.81 to 4.88]

22. Secondary Outcome: Percentage of Participants Satisfied With Study Medication at Week 10
Description: Participants were asked complete the participant Satisfaction with Study Medication question at Week 10 (or early withdrawal). Satisfaction was measured using a single 7-point Likert scale from 1 to 7 where higher scores indicate greater satisfaction with study medication. A score of 1 represents very dissatisfied, whilst a score of 7 represents very satisfied. Participants were categorized as a responder if they are rated either as 6 "Satisfied" or 7 "Very Satisfied". The proportion of responders as percentage of participants based on the participant satisfaction with study medication item was defined as: number of participants with a response of 6 or 7 at the visit divided by number of participants with a satisfaction with study medication assessment at that visit (the sum of responders and non-responders) multiplied by 100.
Time Frame: Week 10
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 145 | 156 | 163
Percentage of participants | 45 | 46 | 64
Statistical Analysis 1: Comparison: Placebo vs GSK372475; Placebo versus GSK372475 in percentage of participants Satisfied with Study Medication at Week 10; Test type: Superiority or Other; p = 0.8782, Regression, Logistic; Odds Ratio (OR) = 0.96, 90% CI 2-sided [0.62 to 1.50]
Statistical Analysis 2: Comparison: Placebo vs Paroxetine; Placebo versus Paroxetine in percentage of participants Satisfied with Study Medication at Week 10; Test type: Superiority or Other; p = 0.0011, Regression, Logistic; Odds Ratio (OR) = 2.45, 90% CI 2-sided [1.56 to 3.86]

23. Secondary Outcome: Number of Participants With Most Severe Suicidal Behaviour and Ideation in the Suicidal Behavior (SB) and Suicidal Ideation (SI) Subscales of the Columbia Suicide Severity Rating Scale (CSSRS) Over Week 10
Description: CSSRS is a clinician-rated scale that evaluates severity and change of suicidality by integrating both behaviour and ideation. For SB scale, participants were scored as "non-suicidal" (00), "preparatory acts or behavior communicating ideation" (01), "aborted attempt" (02), "interrupted attempt" (03) or "actual attempt" (04) based on the most severe score (4 being the most severe). On SI scale, participants were scored as "non-suicidal" (00), "wish to be dead" (01), "non-specific active suicidal thoughts" (02), "active suicidal ideation with associated thoughts of methods without intent" (03), "active suicidal ideation with some intent to act on suicidal thoughts without clear plan" (04), "active suicidal ideation with plan and intent" (05), based on the most severe score (5 being the most severe). For both subscales, 0 indicated absence of symptom and higher score indicated greater severity of symptom. Only those scores for which at least one participant was reported are summarized.
Time Frame: Up to Week 10
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK372475 | Paroxetine
Number analyzed (Participants) | 156 | 171 | 166
Participants
  SB, Score 00, Week 1 | 150 | 168 | 166
  SB, Score 00, Week 2 | 144 | 154 | 154
  SB, Score 00, Week 3 | 139 | 146 | 151
  SB, Score 00, Week 4 | 139 | 140 | 148
  SB, Score 00, Week 5 | 129 | 125 | 141
  SB, Score 00, Week 6 | 132 | 117 | 136
  SB, Score 00, Week 8 | 116 | 105 | 133
  SB, Score 00, Week 10 | 120 | 101 | 130
  SI, Score 00, Week 1 | 130 | 148 | 156
  SI, Score 01, Week 1 | 14 | 17 | 8
  SI, Score 02, Week 1 | 5 | 1 | 1
  SI, Score 03, Week 1 | 1 | 1 | 1
  SI, Score 04, Week 1 | 0 | 1 | 0
  SI, Score 00, Week 2 | 132 | 138 | 148
  SI, Score 01, Week 2 | 7 | 11 | 3
  SI, Score 02, Week 2 | 2 | 4 | 2
  SI, Score 03, Week 2 | 3 | 1 | 1
  SI, Score 04, Week 2 | 0 | 1 | 0
  SI, Score 00, Week 3 | 137 | 135 | 145
  SI, Score 01, Week 3 | 1 | 8 | 4
  SI, Score 02, Week 3 | 1 | 2 | 1
  SI, Score 03, Week 3 | 0 | 1 | 1
  SI, Score 00, Week 4 | 137 | 126 | 143
  SI, Score 01, Week 4 | 1 | 10 | 2
  SI, Score 02, Week 4 | 0 | 4 | 2
  SI, Score 03, Week 4 | 2 | 0 | 1
  SI, Score 00, Week 5 | 123 | 119 | 137
  SI, Score 01, Week 5 | 3 | 5 | 2
  SI, Score 02, Week 5 | 1 | 1 | 1
  SI, Score 03, Week 5 | 3 | 0 | 1
  SI, Score 00, Week 6 | 128 | 112 | 134
  SI, Score 01, Week 6 | 3 | 5 | 1
  SI, Score 02, Week 6 | 0 | 1 | 0
  SI, Score 03, Week 6 | 1 | 0 | 2
  SI, Score 00, Week 8 | 112 | 103 | 130
  SI, Score 01, Week 8 | 3 | 2 | 3
  SI, Score 03, Week 8 | 1 | 0 | 0
  SI, Score 05, Week 8 | 0 | 0 | 1
  SI, Score 00, Week 10 | 118 | 100 | 128
  SI, Score 01, Week 10 | 2 | 1 | 1
  SI, Score 02, Week 10 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to Follow-up (18 weeks).
Description: ITT Population was used.
Arm/Group | Placebo | GSK372475 | Paroxetine
All-Cause Mortality (participants affected / at risk) | 0/156 | 1/171 | 0/166
Serious Adverse Events (participants affected / at risk) | 2/156 | 8/171 | 3/166
Other Adverse Events (participants affected / at risk) | 71/156 | 87/171 | 85/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=156) | GSK372475 (N=171) | Paroxetine (N=166)
Adjustment disorder with mixed disturbance of emotion and conduct (Psychiatric disorders) | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Salpingitis (Infections and infestations) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=156) | GSK372475 (N=171) | Paroxetine (N=166)
Dry mouth (Gastrointestinal disorders) | 4 | 38 | 16
Nausea (Gastrointestinal disorders) | 12 | 18 | 26
Constipation (Gastrointestinal disorders) | 8 | 16 | 14
Diarrhoea (Gastrointestinal disorders) | 9 | 10 | 16
Headache (Nervous system disorders) | 36 | 35 | 26
Somnolence (Nervous system disorders) | 11 | 4 | 17
Dizziness (Nervous system disorders) | 7 | 17 | 7
Insomnia (Psychiatric disorders) | 8 | 17 | 7
Sleep disorder (Psychiatric disorders) | 3 | 10 | 6
Nasopharyngitis (Infections and infestations) | 8 | 5 | 11
Influenza (Infections and infestations) | 6 | 4 | 9
Tachycardia (Cardiac disorders) | 1 | 12 | 3
Palpitations (Cardiac disorders) | 3 | 9 | 3
Fatigue (General disorders) | 8 | 6 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 9 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.